CLINICAL TRIAL: NCT01162681
Title: A Randomized, Double-Blind Phase 2b Study to Evaluate the Efficacy, Safety, and Tolerability of A 623 Administration in Subjects With Systemic Lupus Erythematosus
Brief Title: PEARL-SC Trial: A Study of the Efficacy, Safety, and Tolerability of A 623 Administration in Subjects With Systemic Lupus Erythematosus
Acronym: PEARL-SC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN-SLE3321
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus; Lupus Erythematosus, Systemic; Autoimmune Diseases; A-623; Blisibimod
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — AMG623 peptibody

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A-623 high dose weekly (Experimental)
  Interventions: Drug: A-623
- A-623 low dose weekly (Experimental)
  Interventions: Drug: A-623
- A-623 high dose every 4 weeks (Experimental)
  Interventions: Drug: A-623
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: A-623 — High dose given subcutaneously once a week for up to 52 weeks
  Arms: A-623 high dose weekly
Drug: A-623 — Low dose given subcutaneously once a week for up to 52 weeks
  Arms: A-623 low dose weekly
Drug: A-623 — High dose given subcutaneously once every 4 weeks for up to 52 weeks
  Arms: A-623 high dose every 4 weeks
Other: Placebo Comparator — Placebo comparator is a matched volume given subcutaneously once a week or once every 4 weeks for up to 52 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of three different doses of A-623 administered in addition to standard therapy in subjects with active SLE disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE by American College of Rheumatology guidelines.
* On stable SLE treatment
* Active SLE disease
* Serologically active
* 18 years of age or older
* Receiving stable doses of prednisone between 7.5 mg and 40 mg per day

Exclusion Criteria:

* Severe active vasculitis, active central nervous system lupus, active lupus nephritis, uncontrolled hypertension, or uncontrolled diabetes.
* Known to be positive for HIV and/or positive at the screening visit for hepatitis B, or hepatitis C.
* Liver disease.
* Anemia, neutropenia, or thrombocytopenia.
* Malignancy within past 5 years
* Active infection requiring hospitalization or treatment with parenteral antibiotics within the past 60 days or history of repeated herpetic viral infections.
* History of active tuberculosis or a history of tuberculosis infection.
* Participation in the active treatment arm of any Phase 2 or Phase 3 clinical trial for a molecule that primarily targets the B cell pathway in the past 18 months.
* Prior administration of any B cell depleting therapy in the past 18 months.
* Pregnant or nursing
* History of congenital immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
SLE response | Various timepoints through Week 52
  The % of subjects with SLE response compared with baseline at the time of assessment

SECONDARY OUTCOMES:
B cell reduction | Various timepoints through Week 52
Time to first flare | Various timepoints through Week 52
FACIT-fatigue score | Various timepoints through Week 52
Reduction in prednisone dose | Various timepoints through Week 52
Change in IgG, IgM,C3 and C4 | Various timepoints through Week 52
Flare rates | Various timepoints through Week 52
SRI, using improvements of SELENA-SLEDAI of 5, 6, 7, 8 and 9 | Various timepoints through Week 52

CONTACTS AND LOCATIONS:
Locations (74):
- United States (14):
  - Investigator Site 103, Birmingham, Alabama
  - Investigator Site 113, Long Beach, California
  - Investigator Site 108, Los Angeles, California
  - Investigator Site 110, Upland, California
  - Investigator Site 105, Orlando, Florida
  - Investigator Site 102, Tampa, Florida
  - Investigator Site 117, Baltimore, Maryland
  - Investigator Site 104, Lansing, Michigan
  - Investigator Site 106, Lake Success, New York
  - Investigator Site 114, Smithtown, New York
  - Investigator Site 101, Greenville, North Carolina
  - Investigator Site 112, Oklahoma City, Oklahoma
  - Investigator Site 111, Tulsa, Oklahoma
  - Investigator Site 115, Houston, Texas
- Argentina (7):
  - Investigator Site 404, Caba, Buenos Aires
  - Investigator Site 402, Caba, Buenos Aires
  - Investigator Site 408, San Juan, San Juan Province
  - Investigator Site 403, Rosario, Santa Fe Province
  - Investigator Site 406, San Miguel de Tucumán, Tucumán Province
  - Investigator Site 407, Buenos Aires
  - Investigator Site 401, Buenos Aires
- Brazil (11):
  - Investigator Site 504, Salvador, Estado de Bahia
  - Investigator Site 509, Goiás, Goiania
  - Investigator Site 507, Goiânia, Goiás
  - Investigator Site 506, Juiz de Fora, Minas Gerais
  - Investigator Site 512, Porto Alegre, Rio de Grande Do Sul
  - Investigator Site 503, Rio de Janeiro, Rio de Janeiro
  - Investigator Site 502, Porto Alegre, Rio Grande do Sul
  - Investigator Site 510, Campinas, São Paulo
  - Investigator Site 505, São Paulo, São Paulo
  - Investigator Site 501, São Paulo, São Paulo
  - Investigator Site 511, Rio de Janeiro
- Chile (4):
  - Investigator Site 606, Santiago, Chile
  - Investigator Site 602, Santiago
  - Investigator Site 605, Santiago
  - Investigator Site 601, Viña del Mar
- Colombia (11):
  - Investigator Site 706, Medellín, Antioquia
  - Investigator Site 710, Medellín, Antioquia
  - Investigator Site 701, Barranquilla, Atlántico
  - Investigator Site 704, Barranquilla, Atlántico
  - Investigator Site 703, Bogota, Cundinamarca
  - Investigator Site 707, Bucaramanga, Santander Department
  - Investigator Site 702, Bogotá
  - Investigator Site 705, Bogotá
  - Investigator Site 709, Bogotá
  - Investigator Site 711, Bucaramanga
  - Investigator Site 708, Medellín
- Hong Kong (2):
  - Investigator Site 153, New Territories, Shatin
  - Investigator Site 151, Hong Kong
- India (4):
  - Investigator Site 205, Secunderabad, Andhra Pradesh
  - Investigator Site 203, Bangalore, Kamataka
  - Investigator Site 204, Trivandrum, Kerala
  - Investigator Site 201, Mumbai, Maharashtra
- Mexico (9):
  - Investigator Site 803, Mexico City, D.f.
  - Inestigator Site 809, México, D.f.
  - Investigator Site 806, Guadalajara, Jalisco
  - Investigator Site 804, Morelia, Michoacán
  - Investigator Site 801, San Luis Potosí City, San Luis Potosí
  - Investigator Site 802, Toluca, State of Mexico
  - Investigator Site 808, Guanajuato City
  - Investigator Site 805, México
  - Investigator Site 807, México
- Peru (5):
  - Investigator Site 901, Cayma, Arequipa
  - Investigator Site 903, Lima, Lima Province
  - Investigator Site 905, Lima, Lima Province
  - Investigator Site 904, Lima, Lima Province
  - Investigator Site 902, Bellavista Callao, Provincia Constitucional del Callao
- Philippines (4):
  - Investigator Site 302, Cebu, Cebu
  - Investigator Site 303, Davao City, Davao Region
  - Investigator Site 304, Manila, National Capital Region
  - Investigator Site 305, Davao City
- Taiwan (3):
  - Investigator Site 354, Taichung
  - Investigator Site 352, Taichung
  - Investigator Site 351, Taipei

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Furie RA, Leon G, Thomas M, Petri MA, Chu AD, Hislop C, Martin RS, Scheinberg MA; PEARL-SC Study. A phase 2, randomised, placebo-controlled clinical trial of blisibimod, an inhibitor of B cell activating factor, in patients with moderate-to-severe systemic lupus erythematosus, the PEARL-SC study. Ann Rheum Dis. 2015 Sep;74(9):1667-75. doi: 10.1136/annrheumdis-2013-205144. Epub 2014 Apr 19. PMID 24748629